CLINICAL TRIAL: NCT04923191
Title: Non-inferiority of Angiography-derived Physiology Guidance Versus Usual Care in an All-comers PCI Population Treated With Unrestricted Use of the Healing-Targeted Supreme (HT Supreme) Drug-eluting Stent and P2Y12 Inhibitor Monotherapy After 1-month of Dual-antiplatelet Therapy
Brief Title: The PIONEER-IV Study is Comparing Clinical Outcomes Between Angiography-derived Physiology Guidance to Usual Care in an All-comers PCI Population With Unrestrictive Use of the HT Supreme Sirolimus-eluting Stent
Acronym: PIONEER-IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Patrick Serruys, Professor of Interventional Cardiology & Innovation at the National University of Ireland, Galway, Ireland, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUIG-2021-001
Record Dates: First submitted 2021-06-03; First posted 2021-06-11 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; ischemia; quantitative flow ratio (QFR); P2Y12 monotherapy; drug-eluting stent; physiology guidance; angio-FFR; Coronary Angiography-derived FFR (caFFR)
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography-derived Physiology Guidance: angio-FFR (QFR and caFFR) (Other): Quantitative Flow Ratio- QFR, Coronary angiography-derived FFR - caFFR
  Interventions: Other: Angiography-derived physiology guidance/Local routine diagnostic procedure (LRDP) and usual care
- Local routine diagnostic procedure (LRDP) and usual care (Other)
  Interventions: Other: Angiography-derived physiology guidance/Local routine diagnostic procedure (LRDP) and usual care

INTERVENTIONS:
Other: Angiography-derived physiology guidance/Local routine diagnostic procedure (LRDP) and usual care — percutaneous coronary intervention

SUMMARY:
PIONEER-IV is a prospective, single-blind (patient), randomized, 1:1, controlled, multi-center study comparing clinical outcomes between angiography-derived physiology guidance to LRDP and usual care in an all-comers patient population (including patients with high bleeding risk, HBR) undergoing PCI with unrestrictive use of the HT Supreme sirolimus-eluting stent. Patients will be randomized to either angio-based physiology guidance angio-FFR (Quantitative Flow Ratio and coronary angiography-derived FFR, caFFR) or local routine diagnostic procedure (LRDP) and usual care. Patients will be treated with 1-year P2Y12 inhibitor monotherapy after 1-month of dual-antiplatelet therapy in approximately 2540 (2*1270) patients. All patients (both cohorts) must receive dual anti-platelet therapy, being aspirin (ASA) and ticagrelor for 1 month, followed by 11 months of ticagrelor only (i.e. monotherapy). At 1 year, ticagrelor monotherapy is replaced by aspirin monotherapy or left to the discretion of the operator.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic stable angina, acute coronary syndromes or silent ischemia;
* Presence of one or more coronary artery stenoses of ≥50% (by visual assessment) in a native coronary artery (with or without prior stent/other device treatment) or in a saphenous venous or arterial bypass conduit suitable for coronary stent implantation;
* The vessel should have a reference vessel diameter of at least 2.25 mm by visual assessment (no limitation on the number of treated lesions, vessels, or lesion length);
* Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee and is willing to comply with all protocol-required (follow-up) evaluations.

Exclusion Criteria:

1. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice);
2. Known intolerance to cobalt chromium, and medications such as sirolimus, aspirin, heparin, bivalirudin or P2Y12 inhibitors;
3. Planned major elective surgery requiring discontinuation of (dual)anti platelet therapy (DAPT) within 12 months of procedure;
4. Concurrent medical condition with a life expectancy of less than 3 years;
5. Currently participating in another trial and not yet at its primary endpoint;
6. Active pathological bleeding;
7. History of intracranial haemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2540 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented Composite Endpoint (PoCE) | 12 months
  PoCE is a composite clinical endpoint of:
  * all-cause death;
  * any stroke, Modified Rankin scale, (MRS ≥1);
  * any myocardial infarction;
  * any clinically and physiologically driven revascularization.

SECONDARY OUTCOMES:
Vessel-oriented composite endpoints (VoCE) | 12, 24 and 36 months
  VoCE is a composite clinical endpoint of:
  * Vessel-related cardiovascular Death
  * Target-vessel related MI
  * Clinically and physiologically-oriented Target vessel revascularization
Device-oriented composite endpoint (DoCE) | 12, 24 and 36 months
  DoCE is a composite endpoint of:
  * Cardiovascular Death
  * Target-vessel related MI
  * Clinically and physiologically-oriented Target lesion revascularization
Myocardial Infarction (MI) | 48 hours post-procedure
  Peri-procedure Myocardial Infarction according to 4th universal definition
Device Success Rate | index procedure
  according to the statement from European Association of Percutaneous Cardiovascular Interventions (EAPCI) of the European Society of Cardiology (ESC)
Stent Thrombosis | Procedure, 12, 24 and 36 months
  Definite, Probable, Definite or Probable
Target Vessel Failure (TVF) | 12, 24 and 36 months
  TVF is a composite of:
  * Cardiovascular Death
  * Target-vessel related MI
  * Clinically and physiologically-oriented Target vessel revascularization
Bleeding | 12, 24 and 36 months follow-up
  Bleeding according to Bleeding Academic Research Consortium (BARC) (BARC 2, 3 and 5) classification

CONTACTS AND LOCATIONS:
Locations (19):
- Belgium (5):
  - ASZ Aalst, Aalst
  - OLVZ Aalst, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - CHU Charleroi, Charleroi
  - Jessa Hospital Hasselt, Hasselt
- University Hospital Galway, Galway, Ireland
- Netherlands (6):
  - OLVG Amsterdam, Amsterdam
  - Medisch Spectrum Twente, Thoraxcentrum, Endchede, Enschede
  - UMC Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maasstad Ziekenhuis, Rotterdam
  - Den Haag Ziekenhuis, The Hague
- Spain (4):
  - Hospital Clínico de Barcelona, Barcelona
  - Lucas Augusti Hospital, Lugo
  - Hospital Clínico Universitario of Valladolid, Valladolid
  - Hospital Álvaro Cunqueiro Vigo, Vigo
- United Kingdom (3):
  - Barts Health NHS Trust, London, London
  - Freeman Hospital, Newcastle
  - University Hospitals Southampton, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He X, Tsung-Ying T, Revaiah PC, Wykrzykowska JJ, Rosseel L, Sharif F, Muramatsu T, Reiber JH, Garg S, Miyashita K, Tobe A, Tao L, Onuma Y, Serruys PW. Nomogram based on virtual hyperemic pullback pressure gradients for predicting the suboptimal post-PCI QFR outcome after stent implantation. Int J Cardiovasc Imaging. 2024 Dec;40(12):2469-2479. doi: 10.1007/s10554-024-03253-1. Epub 2024 Oct 12. PMID 39395074
- [Derived] Hara H, Serruys PW, O'Leary N, Gao C, Murray A, Breslin E, Garg S, Bureau C, Reiber JH, Barbato E, Aminian A, Janssens L, Rosseel L, Benit E, Campo G, Guiducci V, Casella G, Santarelli A, Franze A, Diaz VAJ, Iniguez A, Brugaletta S, Sabate M, Amat-Santos IJ, Amoroso G, Wykrzykowska J, von Birgelen C, Somi S, Liu T, Hofma SH, Curzen N, Trillo R, Ocaranza R, Mathur A, Smits PC, Escaned J, Baumbach A, Wijns W, Sharif F, Onuma Y; PIONEER IV trial investigator. Angiography-derived physiology guidance vs usual care in an All-comers PCI population treated with the healing-targeted supreme stent and Ticagrelor monotherapy: PIONEER IV trial design. Am Heart J. 2022 Apr;246:32-43. doi: 10.1016/j.ahj.2021.12.018. Epub 2022 Jan 3. PMID 34990582